CLINICAL TRIAL: NCT01087645
Title: Investigation of Safety, Tolerability and Bioavailability of NN9925 in Healthy Male Subjects
Brief Title: A Two Part Trial Investigating the Safety of NN9925 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9925-3779; 2009-016975-31 (EudraCT Number); U1111-1113-2537 (Other: WHO)
Record Dates: First submitted 2010-03-12; First posted 2010-03-16 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trial part 1 (Experimental)
  Interventions: Drug: NN9925 (oral); Drug: placebo
- Trial part 2 (Experimental)
  Interventions: Drug: NN9925 (i.v.); Drug: NN9925 (oral); Drug: placebo

INTERVENTIONS:
Drug: NN9925 (oral) — Subjects will be randomised to receive a single dose of NN9925, at escalating dose levels. Progression to next dose will be based on safety evaluation
  Arms: Trial part 1
Drug: NN9925 (i.v.) — As an active comparator, one standard dose will be given i.v. (into the vein) at one study visit
  Arms: Trial part 2
Drug: placebo — Subjects will receive a single dose of placebo as a comparator to NN9925, at all dose levels
  Arms: Trial part 1
Drug: NN9925 (oral) — Subjects will be randomised to receive a single dose of NN9925 in up to three different concentrations. The dose will be selected based on the results of part 1
  Arms: Trial part 2
Drug: placebo — Subjects will be randomised to receive a single dose of placebo
  Arms: Trial part 2

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the safety, tolerability and bioavailability (exploring absorption of drug in body) of NN9925 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with good general health as judged by the physician
* Body weight of 65-95 kg (both inclusive)
* Body Mass Index (BMI) of 18.5-27.5 kg/m2 (both inclusive)

Exclusion Criteria:

* Known or suspected allergy to trial product or related products
* Acute infection or inflammation or other illness that may confound the results of the trial or pose a risk to the subject by administering the trial product, as judged by the physician
* Presence of clinically significant acute gastrointestinal symptoms (e.g. nausea, vomiting, heartburn or diarrhoea) or malabsorptive states of disease (celiac disease, lactose intolerance or chronic pancreatitis), as judged by the physician

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2010-03-12 (Actual); Primary Completion 2010-09-16 (Actual); Study Completion 2010-09-16 (Actual)

PRIMARY OUTCOMES:
Number and severity of adverse events (AEs) recorded | from dosing to Day 22

SECONDARY OUTCOMES:
The uptake in blood of oral NN9925 | from 0 to 504 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Nottingham, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com